CLINICAL TRIAL: NCT00083382
Title: UARK 98-036, A Phase II Trial of Combination Bisphosphonate and Anti-Angiogenesis Therapy With Pamidronate and Thalidomide in Patients With Smoldering/Indolent Myeloma
Brief Title: Combination Bisphosphonate and Anti-Angiogenesis Therapy With Pamidronate and Thalidomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-036
Record Dates: First submitted 2004-05-21; First posted 2004-05-24 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Thalidomide; Pamidronate; Aredia; Bisphosphonate; Anti-Angiogenesis; Smoldering/Indolent Myeloma; Zometa
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Pamidronate; Thalidomide; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide + Bisphosphonate (Experimental): 200 mg/day Thalidomide + 90 mg Pamidronate OR 4 mg Zometa every 2 weeks for 2 months and then every 4 weeks as maintenance therapy
  Interventions: Drug: Pamidronate; Drug: Thalidomide; Drug: Zometa

INTERVENTIONS:
Drug: Pamidronate — Patients will receive either pamidronate or zometa. Pamidronate is administered at a dose of 90 mg by continuous infusion over 90 minutes, every two weeks for 2 months. Disease will be reassessed after two cycles. Those with stable disease or better will receive 90 mg every 4 weeks as maintenance therapy.
Drug: Thalidomide — All Patients will receive thalidomide 200 mg as an oral, once daily dose. Dose may be reduced to as low as 50 mg qod in the event of severe toxicity. Thalidomide will continue daily as tolerated until criteria to remove from study are met.
  Patients will receive appropriate regimen to prevent constipation (i.e., colace, dulcolax, milk of magnesia, or lactulose)
Drug: Zometa — Patients will receive either pamidronate or zometa. Zometa is administered at a dose of 4 mg by continuous infusion every two weeks for 2 months. Disease will be reassessed after two cycles. Those with stable disease or better will receive 4 mg every 4 weeks as maintenance therapy.

SUMMARY:
The purpose of this research is to study how helpful the combination of thalidomide and Pamidronate or thalidomide and Zometa is in controlling the myeloma disease and to study any side effects.

DETAILED DESCRIPTION:
Recently laboratory research found that thalidomide can inhibit the formation of new blood vessels that are necessary for the growth and spread of cancer. In order to grow and increase in size tumors require new blood vessels to supply them with the necessary blood to grow. If we can prevent these new blood vessels feeding the tumor from being formed by using thalidomide we might slow or stop the growth of the tumor. This concept is called "anti-angiogenesis" It is hoped that thalidomide will slow or stop the growth myeloma. However, it cannot be guaranteed that you will benefit if you take part in this study. The treatment you receive may even be harmful.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Smoldering or Indolent myeloma
* All patients must be informed of the investigational nature of this study and must sign a written informed consent in accordance with UAMS Human Research Advisory Committee and federal guidelines.

Exclusion Criteria:

* Prior bisphosphonate therapy within 30 days prior to study entry.
* Serum creatinine > 5 mg/dl, ascites, or serum direct bilirubin > 2.5 mg/dl.
* Prior plicamycin or calcitonin within 2 weeks of study entry.
* Severe cardiac disease, unstable thyroid disease, or epilepsy.
* Prior radiation therapy to > 20% of the skeleton.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 1998-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Barlogie B, van Rhee F, Shaughnessy JD Jr, Epstein J, Yaccoby S, Pineda-Roman M, Hollmig K, Alsayed Y, Hoering A, Szymonifka J, Anaissie E, Petty N, Kumar NS, Srivastava G, Jenkins B, Crowley J, Zeldis JB. Seven-year median time to progression with thalidomide for smoldering myeloma: partial response identifies subset requiring earlier salvage therapy for symptomatic disease. Blood. 2008 Oct 15;112(8):3122-5. doi: 10.1182/blood-2008-06-164228. Epub 2008 Jul 31. PMID 18669874
- See also: Myeloma Institute for Research & Therapy — http://myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Thalidomide + Bisphosphonate: 200 mg/day Thalidomide + 90 mg Pamidronate OR 4 mg Zometa every 2 weeks for 2 months and then every 4 weeks as maintenance therapy
  Thalidomide: All Patients will receive thalidomide 200 mg as an oral once daily dose. Dose may be reduced to as low as 50 mg qod in the event of severe toxicity. Thalidomide will continue daily as tolerated until criteria to remove from study are met. Patients will receive appropriate regimen to prevent constipation (i.e., colace, dulcolax, milk of magnesia, or lactulose)
  Pamidronate: Patients will receive either pamidronate or zometa. Pamidronate is administered at a dose of 90 mg by continuous infusion over 90 minutes, every two weeks for 2 months. Disease will be reassessed after two cycles. Those with stable disease or better will receive 90 mg every 4 weeks as maintenance therapy.
  Zometa: Patients will receive either pamidronate or zometa. Zometa is administered at a dose of 4 mg by continuous infusion every two weeks for 2 months. Dise
Period: Overall Study
Arm/Group | Thalidomide + Bisphosphonate
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Thalidomide + Bisphosphonate
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: Best response to study treatment as defined by protocol-specific response criteria:
  Complete Response (CR) = absence of urine and serum M-components by immunofixation; bone marrow should be adequately cellular (>20%) with <1% monoclonal plasma cells by DNA-clg flow cytometry; serum calcium level must be normal; no new bone lesions nor enlargement of existing lesions; Normalization of serum concentrations of normal immunoglobulins is not required for CR. Partial Response (PR) = Reduction by > 75% in serum myeloma protein production; Decrease in monoclonal marrow plasmacytosis to <5%; Decrease in Bence-Jones proteinuria by >90%; No new lytic bone lesions or soft tissue plasmacytoma.
  Treatment Failures/Progressive Disease (PD) = Such patients do not fulfill the above criteria and/or have new lytic lesions (but not compression fractures), hypercalcemia, or other new manifestations of disease.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Thalidomide + Bisphosphonate
Number analyzed (Participants) | 83
participants
  Treatment Failure/Progressive Disease | 56
  Partial Response | 17
  Complete Response | 10

ADVERSE EVENTS:
Arm/Group | Thalidomide + Bisphosphonate
Serious Adverse Events (participants affected / at risk) | 16/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide + Bisphosphonate (N=83)
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Cardiovascular-other (Cardiac disorders) | 3
Joint, muscle, bone-other (Musculoskeletal and connective tissue disorders) | 1
Lung-other (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory infect w/o neutrop (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhea without colostomy (Gastrointestinal disorders) | 1
Fatigue/malaise/lethargy (General disorders) | 1
Syncope (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Speech impairment (General disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
GI-other (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thalidomide + Bisphosphonate (N=83)
Grade 1 Allergic rhinitis (Immune system disorders) | 7
Grade 1 Anemia (Blood and lymphatic system disorders) | 25
Grade 2 Anemia (Blood and lymphatic system disorders) | 8
Grade 1 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 10
Grade 2 Neutropenia/granulocytopenia (Blood and lymphatic system disorders) | 17
Grade 1 Thrombocytopenia (Blood and lymphatic system disorders) | 17
Grade 2 Thrombocytopenia (Blood and lymphatic system disorders) | 5
Grade 3 Thrombocytopenia (Blood and lymphatic system disorders) | 5
Grade 2 Leukopenia (Blood and lymphatic system disorders) | 20
Grade 1 Arrhythmia, NOS (Cardiac disorders) | 9
Grade 4 Cardiovascular - other (Cardiac disorders) | 4
Grade 1 Edema (Cardiac disorders) | 27
Grade 2 Edema (Cardiac disorders) | 8
Grade 1 Hypertension (Cardiac disorders) | 4
Grade 2 Hypertension (Cardiac disorders) | 4
Grade 1 Sinus bradycardia (Cardiac disorders) | 7
Grade 2 Sinus bradycardia (Cardiac disorders) | 5
Grade 1 Fatigue (General disorders) | 23
Grade 2 Fatigue (General disorders) | 42
Grade 3 Fatigue (General disorders) | 9
Grade 1 Fever without neutropenia (General disorders) | 4
Grade 2 Fever without neutropenia (General disorders) | 8
Grade 1 Fever, NOS (General disorders) | 21
Grade 2 Fever, NOS (General disorders) | 12
Grade 2 Sweating (General disorders) | 4
Grade 1 weight gain (General disorders) | 6
Grade 2 weight gain (General disorders) | 5
Grade 1 weight loss (General disorders) | 7
Grade 1 Dry skin (Skin and subcutaneous tissue disorders) | 10
Grade 1 Erythema/rash/eruption/desquamation (Skin and subcutaneous tissue disorders) | 5
Grade 2 Erythema/rash/eruption/desquamation (Skin and subcutaneous tissue disorders) | 9
Grade 1 Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Grade 2 Rash/desquamation (Skin and subcutaneous tissue disorders) | 7
Grade 1 Skin - other (Skin and subcutaneous tissue disorders) | 6
Grade 2 Skin - other (Skin and subcutaneous tissue disorders) | 4
Grade 1 Anorexia (Gastrointestinal disorders) | 9
Grade 2 Anorexia (Gastrointestinal disorders) | 5
Grade 2 Constipation (Gastrointestinal disorders) | 5
Grade 1 Constipation/bowel obstruction (Gastrointestinal disorders) | 24
Grade 2 Constipation/bowel obstruction (Gastrointestinal disorders) | 32
Grade 3 Constipation/bowel obstruction (Gastrointestinal disorders) | 4
Grade 1 Diarrhea without colostomy (Gastrointestinal disorders) | 7
Grade 2 Diarrhea without colostomy (Gastrointestinal disorders) | 9
Grade 1 GI - other (Gastrointestinal disorders) | 7
Grade 1 Mouth dryness (Gastrointestinal disorders) | 12
Grade 2 Mouth dryness (Gastrointestinal disorders) | 9
Grade 1 Nausea (Gastrointestinal disorders) | 11
Grade 2 Nausea (Gastrointestinal disorders) | 8
Grade 1 Vomiting (Gastrointestinal disorders) | 9
Grade 1 Alkaline phosphatase increase (Hepatobiliary disorders) | 4
Grade 1 Hypoalbuminemia (Hepatobiliary disorders) | 36
Grade 2 Hypoalbuminemia (Hepatobiliary disorders) | 7
Grade 1 SGOT (AST) increase (Hepatobiliary disorders) | 12
Grade 1 SGPT (ALT) increase (Hepatobiliary disorders) | 19
Grade 1 Infection w/o 3-4 neutropenia (Infections and infestations) | 6
Grade 2 Infection w/o 3-4 neutropenia (Infections and infestations) | 9
Grade 2 Respiratory infect w/o neutrop (Infections and infestations) | 5
Grade 1 Bicarbonate decrease (Metabolism and nutrition disorders) | 19
Grade 1 Hypercalcemia (Metabolism and nutrition disorders) | 4
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 32
Grade 2 Hyperglycemia (Metabolism and nutrition disorders) | 11
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 6
Grade 1 Hypocalcemia (Metabolism and nutrition disorders) | 39
Grade 2 Hypocalcemia (Metabolism and nutrition disorders) | 9
Grade 1 Hypokalemia (Metabolism and nutrition disorders) | 15
Grade 1 Hypomagnesemia (Metabolism and nutrition disorders) | 47
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 24
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 4
Grade 2 Hypophosphatemia (Metabolism and nutrition disorders) | 22
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 9
Grade 2 Arthritis (Musculoskeletal and connective tissue disorders) | 6
Grade 1 Joint, muscle, bone - other (Musculoskeletal and connective tissue disorders) | 21
Grade 2 Joint, muscle, bone - other (Musculoskeletal and connective tissue disorders) | 16
Grade 3 Joint, muscle, bone - other (Musculoskeletal and connective tissue disorders) | 4
Grade 1 Muscle Weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 11
Grade 2 Muscle Weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 7
Grade 1 Anxiety/agitation (Psychiatric disorders) | 10
Grade 2 Anxiety/agitation (Psychiatric disorders) | 4
Grade 1 Ataxia (Nervous system disorders) | 4
Grade 1 Confusion (Psychiatric disorders) | 13
Grade 2 Confusion (Psychiatric disorders) | 5
Grade 1 Cranial neuropathy (Nervous system disorders) | 6
Grade 1 Depression (Psychiatric disorders) | 19
Grade 2 Depression (Psychiatric disorders) | 11
Grade 1 Dizziness/light headedness (Nervous system disorders) | 14
Grade 2 Dizziness/light headedness (Nervous system disorders) | 5
Grade 3 Dizziness/light headedness (Nervous system disorders) | 7
Grade 1 Headache (General disorders) | 10
Grade 2 Headache (General disorders) | 7
Grade 1 Insomnia (Psychiatric disorders) | 5
Grade 2 Insomnia (Psychiatric disorders) | 5
Grade 1 Memory loss (Psychiatric disorders) | 6
Grade 1 Mood/consciousness change, NOS (Psychiatric disorders) | 9
Grade 1 Neuro - other (Nervous system disorders) | 13
Grade 2 Neuro - other (Nervous system disorders) | 4
Grade 1 Sensory neuropathy (Nervous system disorders) | 39
Grade 2 Sensory neuropathy (Nervous system disorders) | 32
Grade 3 Sensory neuropathy (Nervous system disorders) | 9
Grade 1 Somnolence/consciousness loss (General disorders) | 9
Grade 2 Somnolence/consciousness loss (General disorders) | 5
Grade 3 Somnolence/consciousness loss (General disorders) | 4
Grade 1 Tremor (Nervous system disorders) | 12
Grade 2 Tremor (Nervous system disorders) | 5
Grade 1 Weakness (motor neuropathy) (Nervous system disorders) | 15
Grade 2 Weakness (motor neuropathy) (Nervous system disorders) | 11
Grade 3 Weakness (motor neuropathy) (Nervous system disorders) | 6
Grade 2 Blurred vision (Eye disorders) | 12
Grade 1 Eye - other (Eye disorders) | 8
Grade 1 Bone Pain (General disorders) | 14
Grade 2 Bone Pain (General disorders) | 13
Grade 3 Bone Pain (General disorders) | 6
Grade 1 Chest pain, not cardio or pleural (General disorders) | 4
Grade 2 Lower Back (General disorders) | 4
Grade 1 Pain - other (General disorders) | 10
Grade 2 Pain - other (General disorders) | 10
Grade 3 Pain - other (General disorders) | 5
Grade 1 Upper Back (General disorders) | 6
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 7
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 6
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Grade 3 Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Grade 1 Creatinine increase (Renal and urinary disorders) | 14
Grade 2 Creatinine increase (Renal and urinary disorders) | 5
Grade 1 GU - other (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes